CLINICAL TRIAL: NCT00618085
Title: An Integrated Motor Imagery Program in Rehabilitation - a RCT
Brief Title: Motor Imagery Practice in Neurological Rehabilitation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nuffield Orthopaedic Centre NHS Trust (Other)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Nuffield Orthopaedic Centre NHS Trust, NHS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07/H0605/84NOC; 07/H0605/84
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Stroke; Brain Injury; Multiple Sclerosis
MeSH Terms: conditions — Stroke; Brain Injuries; Multiple Sclerosis | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): All patients will receive the occupational therapy and physiotherapy normally given in their setting.
  In addition; the experimental group will receive 2 instruction DVD's introducing them to motor imagery practice, taking 35 minutes in total. The research therapist will also attend the first session with the physiotherapist and with the occupational therapist to help incorporate motor imagery within the therapy. Thereafter the therapist will help the patient use motor imagery as part of their normal treatment. The total amount spent on motor imagery during therapy sessions will be 6.5 hours in 6 weeks.
  Interventions: Behavioral: Motor imagery practice
- 2 (Active Comparator): All patients will receive the occupational therapy and physiotherapy normally given in their setting.
  In addition; the control group will receive 2 DVDs for 35 minutes in total. These will show background information on their condition, explaining the importance of practice of activities, and on the principles of motor learning and phased movement which underlie most therapy.The research therapist will also attend the first session with the physiotherapist and with the occupational therapist to control for attention. The total amount the physiotherapist and occupational therapist spend with the patients should be the same in both groups.
  Interventions: Other: Standard physiotherapy and occupational therapy

INTERVENTIONS:
Behavioral: Motor imagery practice — During motor imagery practice a person imagines performing a skill or movement with all its sensory consequences without actually moving. In this study the therapists follow a motor imagery guideline designed for rehabilitation of skills and movement performance in subjects with neurological disease or damage. The guideline offers therapists structure and a strategy to deliver subject-specific imagery. The guideline is based on three major frameworks, namely; principles of motor learning, phased process of human movement and a training guide for sports coaches and performers from the National Coaching Foundation.
  Arms: 1
Other: Standard physiotherapy and occupational therapy — Patients with neurological disease or damage will receive standard physiotherapy and occupational therapy.
  Arms: 2

SUMMARY:
Motor imagery is a technique widely used in learning skills. Its effectiveness has been proven in various sports and in musicians. A recent review (Braun et al. 2006) suggested that this technique may also be effective in rehabilitation of patients with neurological disease or damage, but that further research was needed.

The main purpose of this research is to discover whether motor imagery practice is beneficial in the rehabilitation of skills in patients who have some disability due to neurological disease or damage. The principal research question is: are physiotherapy and occupational therapy given incorporating motor imagery more effective than standard care (i.e., the same therapies but without integrated motor imagery) in re-training task specific performance for patients with neurological disease or damage?

ELIGIBILITY:
Inclusion Criteria:

* Participating in a rehabilitation program for problems arising secondary to disease or damage affecting the central nervous system (usually stroke, brain injury, multiple sclerosis)
* Over 18 years of age
* Have sufficient language and memory skills to undertake the intervention (i.e. score positive on the first three items of the Sheffield screening test)

Exclusion Criteria:

* Any co-morbidity that would interfere with the ability to perform imagery as judged by the clinician or from the medical notes (e.g., schizophrenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scaling | After 6 and 12 weeks

SECONDARY OUTCOMES:
Motor imagery questionnaire | Baseline, 6 weeks, 12 weeks
Timed up and go | Baseline, 6 weeks, 12 weeks
Action research arm test | Baseline, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thamar J Bovend'Eerdt, MSc, Principal Investigator — Oxford Centre for Enablement; Derick T Wade, MD, Study Director — Oxford Centre for Enablement
Locations (1):
- Oxford Centre for Enablement, Oxford, United Kingdom

REFERENCES:
- [Background] Braun SM, Beurskens AJ, Borm PJ, Schack T, Wade DT. The effects of mental practice in stroke rehabilitation: a systematic review. Arch Phys Med Rehabil. 2006 Jun;87(6):842-52. doi: 10.1016/j.apmr.2006.02.034. PMID 16731221